CLINICAL TRIAL: NCT00657670
Title: Evaluation of the Feasibility of Correcting Refractive Error From a Limited Inventory of Ready-made Spectacles: Wearer Retention, Vision Function, Quality of Life and Cost
Brief Title: Evaluation of Effectiveness of Correcting Refractive Error With Ready-made Spectacles
Acronym: RECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Lisa Keay, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA00013454
Record Dates: First submitted 2008-04-11; First posted 2008-04-14 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Myopia; Hyperopia; Astigmatism
Keywords: refractive error; spectacles; ready made spectacles; vision; cost effectiveness
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ready-made spectacles
  Interventions: Device: Ready-made spectacles
- 2 (Active Comparator): Spectacles
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Ready-made spectacles — Ready-made spectacles will be dispensed to correct refractive error. Ready-made spectacles are spectacles which are available from an existing inventory. This is different to prescription spectacles which are usually made to order. They have the same spherical power for the right and left eyes and do not include a correction for astigmatism. The limited inventory for this trial includes +1.00 to +4.00 in 0.50 steps, +5.00, +6.00 and +8.00, -1.00 to -6.00 in 0.50 steps, -7.00, -8.00, -9.00 and -10.00. The appropriate spectacles are selected based on the spherical equivalent refractive error. If there is a difference between the two eyes the lower correction is selected.
  Other Names: Off-the-shelf spectacles
  Arms: 1
Device: Spectacles — Spectacles will be prescribed to correct refractive error. These spectacles will be custom-prescribed based on the sphero-cylindrical refractive correction. The spectacles used in this arm will be custom made for each participant based on their refraction and can be made in a full range of spherical powers and astigmatic corrections for up to 2.00 dioptres of cylinder.
  Other Names: Prescription glasses
  Arms: 2

SUMMARY:
This research project will compare two methods of correcting refractive error (long or short-sightedness) with spectacle lenses. The primary outcome is the proportion of the population requiring spectacle correction who's needs are met through each scheme. Secondary outcomes are the cost effectiveness of these schemes and development of guidelines for identification of those amongst the population suitable for 'ready-made' spectacles.

There are two sites involved in this research. Those with uncorrected refractive error will be identified by their distance vision. Those who have impaired vision (at least 20/40) which improves with spectacles will be invited to participate in this research. Participants will be randomly allocated to one of two groups. The first group will receive spectacles with full correction in both eyes and the second group will receive spectacles from a limited inventory. The two schemes will be compared by how many people continue to use the spectacles, vision with the new spectacles, change in the level of visual functioning and quality of life after wearing new spectacles for one month. At the one month visit, if the spectacles provided are not useful, one new pair of custom spectacles will be dispensed.

DETAILED DESCRIPTION:
In India, participants will be recruited from those attending Shroff's Charity Eye Hospital for refractive eye care. These individuals are screened for eye disease and visual acuity is measured as part of routine care. All with distance vision worse than 20/40 will have pinhole acuity taken to estimate benefit of refractive correction. Those who have refracted distance visual acuity better than 20/40 in the better eye and minimum spherical refractive error of ±1 dioptre will be eligible for the study. The clinical testing can be conducted on the same day and include habitual distance vision, refraction and refracted visual acuity.

In China, participants will be recruited from those identified by a School Screening Program in place in GuangZhou (Childsight). In this program, teachers measure visual acuity. Those who have 20/40 or worse distance vision will be invited to a parent information night. At this time, information will be provided about the study and those interested in participating will sign a record of informed assent with parental permission. The clinical testing will be conducted at a later visit by an optometrist attending the school. Study questionnaires will be administered and clinical testing of vision including habitual distance vision, refraction and refracted visual acuity.

The duration of the study will be up to 2 months and will require a total of three visits. After the initial visit, the dispensing visit will be arranged based on time to supply spectacles and the final visit planned for 1 month after receipt of spectacles.

This study will be masked. The persons interviewing the patients about quality of life and those testing vision on both visits will not know the intervention status of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Presenting visual acuity of 20/40 or worse in the better eye, who have improvement to 20/40 or better following refraction
* A minimum of 1 dioptre of spherical refractive error must be present
* Aged 18-45 years of age at Shroffs Charity Eye Hospital
* Junior High School Students approximate age 11-16 years of age at Zhongshan Ophthalmic Center

Exclusion Criteria:

* Those who do not correct to within 20/40 with spectacle correction.

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Wearer retention (% wearing at 1 month), vision (logMAR), visual function (0-100), quality of life (0-100) | a 1-month period of spectacle wear

SECONDARY OUTCOMES:
Cost-effectiveness | 1-month of spectacle wear
Willingness to pay | 1-month of spectacle wear
Recommendations for those who will benefit from ready made spectacles | 1-month of spectacle wear
Quantify the prismatic effects which has an impact of spectacle compliance, need for adaptation and satisfaction with spectacles | 1-month of spectacle wear
Continued spectacle use 6-12 months after dispensing | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Keay, PhD BOptom, Principal Investigator — Johns Hopkins University; Guofu Huang, MD, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Monica Gandhi, MD, Study Director — Shroffs Charity Eye Hospital
Locations (2):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China
- Shroffs Charity Eye Hospital, New Delhi, India

REFERENCES:
- [Result] Zeng Y, Keay L, He M, Mai J, Munoz B, Brady C, Friedman DS. A randomized, clinical trial evaluating ready-made and custom spectacles delivered via a school-based screening program in China. Ophthalmology. 2009 Oct;116(10):1839-45. doi: 10.1016/j.ophtha.2009.04.004. Epub 2009 Jul 9. PMID 19592103
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Angell B, Ali F, Gandhi M, Mathur U, Friedman DS, Jan S, Keay L. Ready-made and custom-made eyeglasses in India: a cost-effectiveness analysis of a randomised controlled trial. BMJ Open Ophthalmol. 2018 Feb 9;3(1):e000123. doi: 10.1136/bmjophth-2017-000123. eCollection 2018. PMID 29657979